CLINICAL TRIAL: NCT03718962
Title: The Effect of UVB Phototherapy With Microneedling and Circled Needing in Vitiligo Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180205R
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-12

CONDITIONS: Brief Description of Focus of Study Instead
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- needling (Active Comparator): needling + phototherapy
  Interventions: Device: Surrounding needling+ phototherapy
- phototherapy (Placebo Comparator): phototherapy
  Interventions: Device: phototherapy

INTERVENTIONS:
Device: Surrounding needling+ phototherapy — Surrounding needling+ phototherapy
  Other Names: phototherapy
  Arms: needling
Device: phototherapy — phototherapy
  Arms: phototherapy

SUMMARY:
Vitiligo is a relatively common acquired disorder of pigmentation characterized by the development of well-defined white macules on the skin. Biopsies of lesional skin reveal a loss of epidermal melanocytes. Lesions may occur in a localized or generalized distribution and may coalesce into large, depigmented areas. Given the contrast between the white areas and normal skin, the disease is most disfiguring in darker skin types and has a profound impact on the quality of life of both children and adults . Patients with vitiligo often experience stigmatization, social isolation, and low self-esteem. The therapys include topical steroids, topical immunosuppresant, systemic steroids, phototherapy, and surgery.

The aim of this study is to investigate the effect of phototherpy and accupuncture combined therapy for vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Vitiligo

Exclusion Criteria:

* pregnancy
* immune disorder
* infection
* other dermatosis in treating areas

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
repigmentation | 12weeks
  repigmentation amount

CONTACTS AND LOCATIONS:
Locations (1):
- ShinKongHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No